CLINICAL TRIAL: NCT00294996
Title: A Phase III Randomized, Controlled Trial of Myocet, Trastuzumab and Paclitaxel Versus Trastuzumab and Paclitaxel for First-Line Therapy of Metastatic Breast Cancer
Brief Title: Trial of Myocet in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sopherion Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STM01-102
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer
Keywords: Metastatic Her2+ Breast cancer; Myocet; liposomal doxorubicin; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin

INTERVENTIONS:
Drug: Myocet

SUMMARY:
The purpose of the study is to examine the safety and effectiveness of the drug combination of Myocet, paclitaxel and trastuzumab compared to paclitaxel and trastuzumab without Myocet, as first line treatment for patients with metastatic HER2+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic Her2+ Breast cancer by FISH analysis
* No prior chemotherapy for metastatic disease
* Measurable disease
* normal left ventricular ejection fraction

Exclusion Criteria:

* prior doxorubicin treatment exceeding 300 mg/m2 or epirubicin exceeding 600 mg/m2
* relapse within 12 months of completion of adjuvant trastuzumab, taxane or anthracycline therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2006-01

PRIMARY OUTCOMES:
Progression-Free Survival

SECONDARY OUTCOMES:
Overall Survival
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Jose Baselga, M.D., Principal Investigator — Vall d'Hebron Hospital, Barcelona, Spain
Locations (105):
- United States (18):
  - Scripps Cancer Center Clinical Research, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Northwest Hematology/Oncology Associates, Coral Springs, Florida
  - Osceola Cancer Center, Kissimmee, Florida
  - UM/Sylvester Cancer Center, Plantation, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Clintell, Inc, Skokie, Illinois
  - Hutchinson Clinic P.A., Hutchinson, Kansas
  - Western Maryland Health System, Cumberland, Maryland
  - Brody School of Medicine @ ECU, Greenville, North Carolina
  - Aultman Hospital Cancer Center, Canton, Ohio
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - Vita Hematology Oncology, Bethlehem, Pennsylvania
  - Hematology & Oncology Associates of NEPA, Dunmore, Pennsylvania
  - PA Oncology Hematology Asso, Philadelphia, Pennsylvania
  - M. Francisco Gonzalez, Columbia, South Carolina
  - Sioux Valley Clinic, Sioux Falls, South Dakota
  - Tennessee Cancer Specialists, Knoxville, Tennessee
- Argentina (10):
  - Centro Oncologico de Excelencia, Buenos Aires
  - Hospital Enrique Tornú, Buenos Aires
  - Hospital Interzonal Gral de Agudos " EVITA", Buenos Aires
  - Hospital Profesor A. Posadas, Buenos Aires
  - Santorio Municipal Dr. J. Mendez, Buenos Aires
  - Unidad Oncologica del Neuquen, Neuquén
  - CAICI Instituto, Santa Fe
  - Centro Oncologico Rosario, Santa Fe
  - ISIS Clinica Especializada, Santa Fe
  - Ceten, Villa Domínico
- Canada (10):
  - Dr. Leon Richard Oncology Centre, Moncton, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - London Regional Cancer Centre/London Health Science Centre, London, Ontario
  - The Ottawa Hospital Regional Cancer Center, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUM Hospital Notre-Dame, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Hopital du St. Sacrement, Québec
- Germany (7):
  - U.K Charité, Campus Mitte, Berlin
  - Universitätsklinikum Magdeburg, Magdeburg
  - Gemeinschaftspraxis Gynäkologie & Geburtshilfe, Mannheim
  - Frauenklinik von Roten Kreuz, München
  - Klinikum Offenbach, Offenbach
  - Üniversitäts Klinikum Tübingen, Tübingen
  - Dr. Horst Schmidt Kliniken, Wiesbaden
- India (17):
  - Gujarat Cancer Research Institute, Asarwa, Gujarat
  - Kidwai Memorial Institute of Oncology, Bangalore
  - Manipal Hospital, Bangalore
  - Apollo Specialty Hospitals, Chennai, Chennai
  - Nizam's Institute of Medical Science, Hyderabaad
  - SMSMedicalCollegeHospital,, Jaipur
  - Lakeshore Hospital and Research Centre Ltd, Kerala
  - Himadri cancer welfare trusr, Kolkata
  - Orchid Nursing Home,, Kolkata
  - Ruby Hall Clinic, Maharashtra
  - Tata Memorial Hospital, Maharashtra
  - Kasturba Medical College,, Mangalore
  - Jaslok Hospital and Research Centre, Mumbai
  - Batra Hospital & Medical Research Center, New Delhi
  - Indraprastha Apollo Hospitals, New Delhi
  - Safdarjung Hospital & Vardhaman Mahaveer Medical College, New Delhi
  - Fortis Hospital, Noida
- Italy (7):
  - Azienda Ospedialera Pugliese-Ciaccio, Catanzaro
  - Clinica Oncologica Ospedale, Chieti
  - DIMI - Università di Genova, Genova
  - ARNAS CIVICO. Presidio Ospedaliero M. Ascoli, Palermo
  - Oncologia Medica, Pavia
  - Day Hospital Oncologico,, Roma
  - Istituto Clinico Humanitas, Rozzano
- Poland (10):
  - SP SK nr1 ACK AMG, Gdansk
  - Centrum Onkologii - Instytut Marii Skłodowskiej-Curie Oddział Gliwice, Gliwice
  - Regionalny Ośrodek Onkologiczny, Lodz
  - Samodzielny Publiczny Szpital, Lublin
  - Zakład Opieki Zdrowotnej MSWiA, Olsztyn
  - Regionalny Szpital Specjalistyczny, Swidnica
  - Szpital Wojewódzki im. Św. Łukasza, Tarnów
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - SP ZOZ Szpital Wojewódzki, Zielona Góra
- nstituto Português de Oncologia Francisco Gentil, Lisbon, Portugal
- Russia (10):
  - Non-state Health Care Insitution "N.A. Semashko Central Clinical Hospital #2" of the "Russian Railways" Joint Stock Company, Moscow
  - State Institution "N.N. Blokhin Russian Oncology Scientific Center" of the Russian Academy of Medical Sciences, Moscow
  - State Science Institution "P.A. Hertzen Moscow Oncology Research Institute" of the Federal Agency of Health Care and Social Development, Moscow
  - State Health Care Institution "Regional Clinical Oncology Dispensary", Ryazan
  - Research Institute of Pulmonology affiliated with State Educational Institution "St. Petersburg State Medical University n.a. academician I.P. Pavlov" of the Federal Agency of Health Care and Social Development, Saint Petersberg
  - St. Petersburg State Health Care Institution "City Clinical Oncology Dispensary", Saint Petersberg
  - State Science Institution "Prof. N.N. Petrov Research Institute of Oncology" of the Federal Agency of Health Care and Social Development, Saint Petersberg
  - State Health Care Institution "Leningrad Regional Oncology Dispensary", Saint Petersburg
  - Municipal Health Care Institution of the City of Sochi "Oncology Dispensary", Sochi
  - State Health Care Institution of the Yaroslavl Region "Yaroslavl Regional Oncology Dispensary", Yaroslavl
- Spain (11):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital 12 de Octubre, Madrid
  - Hospital Son Dureta, Palma de Mallorca
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Virgen Macarena, Seville
  - Hospital Mutua de Terrassa, Terrassa
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- United Kingdom (4):
  - Broomfield Hospital, Broomfield
  - Christie Hospital NHS Trust, Cardiff
  - Guy's Hospital, London
  - Royal Free Hospital, London

REFERENCES:
- [Derived] Baselga J, Manikhas A, Cortes J, Llombart A, Roman L, Semiglazov VF, Byakhov M, Lokanatha D, Forenza S, Goldfarb RH, Matera J, Azarnia N, Hudis CA, Rozencweig M. Phase III trial of nonpegylated liposomal doxorubicin in combination with trastuzumab and paclitaxel in HER2-positive metastatic breast cancer. Ann Oncol. 2014 Mar;25(3):592-598. doi: 10.1093/annonc/mdt543. Epub 2014 Jan 8. PMID 24401928